CLINICAL TRIAL: NCT02865343
Title: Ventilatory Support to Improve Exercise Training in High Level Spinal Cord Injury
Acronym: NIV-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, Principle Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P000658
Record Dates: First submitted 2016-07-15; First posted 2016-08-12 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Injury
Keywords: Functional Electrical Stimulation (FES)-Rowing
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and technicians helping for performing the test and encouraging the patient will be blind. Only one investigator will monitor the ventilation during the test and won't be blind but won't be participating to any encouragement or data acquisition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Non-invasive Ventilation(NIV) (Active Comparator): Subjects randomized to NIV will perform 12-weeks of FES-row training while receiving bi-level positive airway pressure ventilation applied through a full face-mask.
  Interventions: Device: Non-invasive Ventilation(NIV)
- Sham Non-invasive ventilation(NIV) (Placebo Comparator): Subjects randomized to Sham-NIV will perform 12-weeks of FES-row training while receiving sham ventilation applied through a full face-mask.
  Interventions: Device: Sham Non-invasive ventilation(NIV)

INTERVENTIONS:
Device: Non-invasive Ventilation(NIV) — The ventilator will be set in spontaneous mode with a ramp to reach a minimal pressure of 12 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Arms: Non-invasive Ventilation(NIV)
Device: Sham Non-invasive ventilation(NIV) — The ventilator will be set in spontaneous mode with a ramp to reach a maximal pressure of 5 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Arms: Sham Non-invasive ventilation(NIV)

SUMMARY:
The investigators have an existing exercise program (N>70) with a unique population of individuals with spinal cord injury (SCI) who have been enrolled in FES-RT for at least 6 months. Roughly half have high level SCI. Thirty individuals with high level SCI who have FES-row trained for at least 6 months will be randomized to (continued) FES-RT for 3 months with either NIV or sham NIV. Before and after training, the investigators will assess maximal aerobic capacity, ventilation, cardiac output, and arterio-venous oxygen difference. Based on the investigators current data, it is hypothesized that only those randomized to NIV will experience further increases in aerobic capacity and that these increases will relate to increases in cardiac output and arterio-venous oxygen difference. This Exploratory/Developmental Research project will lay the groundwork for a larger study of the impact of FES-RT+NIV to improve health and function in those with high level SCI.

DETAILED DESCRIPTION:
Regular aerobic exercise with sufficient intensity can improve overall health, however daily energy expenditure is low in those with SCI, especially in those with high level lesions. We have developed Functional Electrical Stimulation Row Training (FESRT) that couples volitional arm and electrically controlled leg exercise, increasing the active muscle and resulting in benefits of large muscle mass exercise. Despite the potential for enhancing aerobic capacity, those with high level lesions (C4 to T2) have a remaining obstacle to attaining higher work capacities they have the greatest pulmonary muscle denervation and our preliminary work suggests this limits the aerobic capacity that can be achieved with FESRT. External ventilatory support could improve the ability to exercise train and hence enhance the adaptations to chronic exercise in high level SCI. Non invasive ventilation (NIV) during exercise training has been shown to improve gains in exercise capacity in those with similarly restrictive breathing. Therefore, the investigators hypothesize that the use of NIV during FESRT will reduce ventilatory limits to exercise, leading to increased aerobic capacity in high level SCI. Our aims are to determine the magnitude of improvement in aerobic capacity and its relationship to increases in maximal cardiac output and arterio venous oxygen difference after 3 months of FESRT+NIV compared to FESRT+shamNIV. The investigators have access to a large (N>70) and unique population of individuals with SCI who have been enrolled in FESRT for at least 6 months. Roughly half have SCI between C4 and T2. 30 individuals with high level SCI who have FES row trained for at least 6 months will be randomized to (continued) FESRT for 3 months with either NIV or sham NIV. Before and after training, the investigators will assess maximal aerobic capacity, ventilation, cardiac output, and arterio venous oxygen difference. Based on our current data, it is hypothesized that only those randomized to NIV will experience further increases in aerobic capacity and that these increases will relate to increased cardiac output and arterio venous oxygen difference. This Exploratory/Developmental Research project will determine feasibility and effectiveness of this approach to exercise and will lay the groundwork for a larger, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 60
* Have had high level SCI (neurological level ≥T3 with American Spinal Injury Association grade A or B or C)
* Medically stable
* Have FES-row trained for >6 months

Exclusion Criteria:

* Hypertension(Blood pressure>140/90 mmHg)
* Significant arrhythmias
* Coronary disease
* Chronic respiratory disease
* Diabetes
* Renal disease
* Cancer
* Epilepsy
* Current use of cardioactive medications
* Current grade 2 or greater pressure ulcers at relevant contact sites
* Other neurological disease
* Peripheral nerve compression or rotator cuff tears that limit the ability to row
* History of bleeding disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vivodtzev I, Picard G, Cepeda FX, Taylor JA. Acute Ventilatory Support During Whole-Body Hybrid Rowing in Patients With High-Level Spinal Cord Injury: A Randomized Controlled Crossover Trial. Chest. 2020 May;157(5):1230-1240. doi: 10.1016/j.chest.2019.10.044. Epub 2019 Nov 16. PMID 31738927

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-invasive Ventilation(NIV) | Sham Non-invasive Ventilation(NIV)
Started | 6 | 5
Completed | 6 | 3
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-invasive Ventilation(NIV) | Sham Non-invasive Ventilation(NIV) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (15) | 31 (8) | 39 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Aerobic Capacity After 3 Months of FES-row Training.
Description: Volunteers will perform a maximal incremental FES-row tests. Both NIV Support and Sham-NIV groups will perform tests in the Sham-NIV condition
Time Frame: Baseline and 3 months
Population: Only participants who reached the criteria of maximality during the maximal incremental test
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Non-invasive Ventilation(NIV) | Sham Non-invasive Ventilation(NIV)
Number analyzed (Participants) | 3 | 3
L/min | 0.21 (0.04) | 0.08 (0.10)

2. Secondary Outcome: Change in Peak Cardiac Output After 3 Months of FES-row Training.
Description: as for outcome 1
Time Frame: Baseline and 3 months
Population: only individuals who sustained exercise while measuring CO
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Non-invasive Ventilation(NIV) | Sham Non-invasive Ventilation(NIV)
Number analyzed (Participants) | 1 | 2
L/min | 2.8 (0) | -2.2 (1.8)

3. Secondary Outcome: Change in Baseline Peak Minute Ventilation During Exercise After 3 Months of FES-row Training
Description: as for outcome 1
Time Frame: Baseline and 3 months
Population: Only individuals who reached maximality during the maximal incremental test
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Non-invasive Ventilation(NIV) | Sham Non-invasive Ventilation(NIV)
Number analyzed (Participants) | 3 | 3
L/min | 1.4 (2.1) | 3.1 (1.6)

ADVERSE EVENTS:
Time Frame: 3 months
Description: This study was investigating the effect of an additional tool during exercise training to increase aerobic capacity during exercise. Adverse events has been collected during the whole period of the study.
Arm/Group | Non-invasive Ventilation(NIV) | Sham Non-invasive Ventilation(NIV)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
The repeatability of maximal exercise tests is difficult in Spinal cord injury, increasing variability of measures an limiting data availability. Higher number of participants will be necessary to study the effect of NIV on the aerobic capacity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02865343/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT02865343/ICF_001.pdf